CLINICAL TRIAL: NCT01049633
Title: B-Lymphocyte Immunotherapy in Islet Transplantation: Single Subject Modification to Calcineurin-Inhibitor Based Immunosuppression for Initial Islet Graft (CIT-0501)
Brief Title: B-Lymphocyte Immunotherapy in Islet Transplantation for Initial Islet Graft Failure
Status: No longer available | Type: Expanded Access
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: DAIT CIT-0501
Record Dates: First submitted 2010-01-12; First posted 2010-01-14 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Insulin dependence; Hypoglycemia; Hypoglycemia unawareness; Islet transplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Sirolimus; Basiliximab; Tacrolimus; Anti-Infective Agents; Antifungal Agents; Trimethoprim, Sulfamethoxazole Drug Combination; Clotrimazole; Valganciclovir; Heparin; Enoxaparin; Pentoxifylline; Aspirin

INTERVENTIONS:
Biological: Allogeneic Pancreatic Islet Cells — 200mL sterile suspension of allogeneic human pancreatic islets
Drug: Sirolimus — Dosed to maintain whole blood 24-hr trough levels 10-15ng/mL for first 3 months and 8-12ng/mL thereafter daily. Sirolimus is used to prevent transplant rejection.
Biological: Basiliximab — 20mg intravenously (IV) 2hrs prior to islet infusion and on Day 4 post-transplant. Basiliximab is used to prevent transplant rejection
Drug: Tacrolimus — Initial dose of 0.015mg/kg p.o. daily on Day 1 post transplant, and adjusted to maintain 12-hr trough levels 3-6ng/mL. Tacrolimus lowers the risk of organ rejection
Drug: Antibacterial, Antifungal, and Antiviral Prophylaxis — Broad spectrum antimicrobial prophylaxis administered preoperatively
Drug: Trimethoprim/sulfamethoxazole — 80mg/400mg by mouth once a day starting on Day 1 for duration of the study follow-up. This medication is used to prevent bacterial infections.
  Other Names: Septra SS
Drug: Clotrimazole — 1 troche by mouth 4 times daily starting two days prior to transplant until 3 months after the transplant. This medication is used to prevent fungal infections.
  Other Names: Mycelex Troche
Drug: Valganciclovir — 450mg dose by mouth once a day starting two days pre-transplant and increasing to 900 mg once a day by Day 12 and continuing for 14 weeks post-transplant. This medication is used to prevent cytomegalovirus infections.
  Other Names: Valcyte
Drug: Heparin — 70U/kg body weight of recipient given with islet infusion, followed by 3U/kg/hr for the next 4hrs. From 5th through 48th hr post-transplant heparin will be titrated to achieve and maintain a Partial Thromboplastin Time (PTT) of 50-60 seconds. This medication is used to prevent the formation of blood clots.
  Other Names: Anticoagulation and Hematological Agent
Drug: Enoxaparin — 30mg subcutaneously twice a day from 48 hrs post-transplant through Day 7 post-transplant. This medication is used to prevent the formation of blood clots.
  Other Names: Lovenox; Anticoagulation and Hematological Agent
Drug: Pentoxifylline — 400mg slow release tablet by mouth three times a day beginning 2 days prior to transplant and continue for 7 days post transplant. This medication improves blood flow.
  Other Names: Anticoagulation and Hematological Agent
Drug: Aspirin — 81mg enteric coated aspirin by mouth every night, starting 24hrs post-transplant. This medication prevents blood clots.
  Other Names: ASA; Anticoagulation and Hematological Agent

SUMMARY:
Type 1 diabetes is an autoimmune disease in which the insulin-producing pancreatic beta cells are destroyed, resulting in poor blood sugar control. The purpose of this study is to determine the safety and effectiveness of islet transplantation, combined with immunosuppressive medications and medications to support islet survival for treating type 1 diabetes in individuals experiencing hypoglycemia unawareness and severe hypoglycemic episodes.

DETAILED DESCRIPTION:
Type 1 diabetes is commonly treated with the administration of insulin, either by multiple insulin injections or by a continuous supply of insulin through a wearable pump. Insulin therapy allows long-term survival in individuals with type 1 diabetes; however, it does not guarantee constant normal blood sugar control. Because of this, long-term type 1 diabetic survivors often develop vascular complications, such as diabetic retinopathy, an eye disease that can cause poor vision and blindness, and diabetic nephropathy, a kidney disease that can lead to kidney failure. Some individuals with type 1 diabetes develop hypoglycemia unawareness, a life-threatening condition that is not easily treatable with medication and is characterized by reduced or absent warning signals for hypoglycemia. For such individuals, pancreas or pancreatic islet transplantation are possible treatment options. Insulin independence among islet transplant recipients tends to decline over time. New strategies aimed at promoting engraftment of transplanted islets are needed to improve the clinical outcomes associated with this procedure.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in clinical trial DAIT CIT-05 (NCT00468442)
* Islet graft failure: absent stimulated C-peptide (<0.3ng/mL) in response to mixed meal tolerance test

Exclusion Criteria:

* Untreated proliferative diabetic retinopathy
* Blood Pressure: systolic blood pressure>160mmHg or diastolic blood pressure>100mmHg
* Measured glomerular filtration rate (GFR) using iohexol < 80ml/min/1.73m^2 Strict vegetarians with a calculated GFR < 70ml/min/1.73m^2
* Presence or history of macroalbuminuria > 300mg/g of creatinine
* Presence or history of panel-reactive anti-HLA antibodies above background by flow cytometry
* For female participants: Positive Pregnancy Test, presently breast-feeding, or unwillingness to use effective contraceptive measures for the duration of the study and 3 months after discontinuation. For male participants: intent to procreate during the duration of the study or within 3 months after discontinuation or unwillingness to use effective measures of contraception. Oral contraceptives, Norplant, Depo-Provera and barrier devices with spermicide are acceptable contraceptive methods; condoms used alone are not acceptable.
* Active infection including hepatitis B, hepatitis C, HIV, or TB as determined by a positive skin test or clinical presentation, or under treatment for suspected TB. Positive tests are acceptable only if associated with a history of previous vaccination in the absence of any sign of active infection. Positive tests are otherwise not acceptable, even in the absence of any active infection at the time of evaluation.
* Negative screen for Epstein-Barr Virus (EBV) by IgG determination
* Invasive aspergillus, histoplasmosis, or coccidiomycosis infection within one year prior to study enrollment
* Any history of malignancy except for completely resected squamous or basal cell carcinoma of the skin
* Known active alcohol or substance abuse
* Anemia (Hgb < 11 g/dL),neutropenia (<1,500/µL), or thrombocytopenia (platelets <100,000/µL)
* A history of Factor V deficiency
* Any coagulopathy or medical condition requiring long-term anticoagulant therapy (e.g., warfarin) after transplantation (low-dose aspirin treatment is allowed) or patients with an International Normalized Ratio (INR) >1.5
* Severe co-existing cardiac disease, characterized by any one of these conditions:

  1. recent myocardial infarction (within past 6 months)
  2. evidence of ischemia on functional cardiac exam within the last year
  3. left ventricular ejection fraction <30%
* Persistent elevation of liver function tests (LFTs) at the time of study entry (e.g., persistent SGOT (AST), SGPT (ALT), Alk Phos or total bilirubin, with values >1.5 times normal upper limits
* Symptomatic cholecystolithiasis
* Acute or chronic pancreatitis
* Symptomatic peptic ulcer disease
* Severe unremitting diarrhea, vomiting or other gastrointestinal disorders potentially interfering with the ability to absorb oral medications
* Hyperlipidemia despite medical therapy (fasting LDL cholesterol > 130 mg/dL, treated or untreated; and/or fasting triglycerides > 200 mg/dL)
* Receiving treatment for a medical condition requiring chronic use of systemic steroids, except for the use of ≤ 5 mg prednisone daily, or an equivalent dose of hydrocortisone, for physiological replacement only
* Use of any investigational agents within 4 weeks of enrollment
* Administration of live attenuated vaccine(s) within 2 months of enrollment
* Any medical condition that, in the opinion of the investigator, will interfere with the safe completion of the trial, such as chronic central neurologic disease
* Treatment with any anti-diabetic medication other than insulin within 4 weeks of enrollment
* A previous pancreas transplant, unless the graft failed within the first week due to thrombosis, followed by pancreatectomy and the transplant occurred more that 6 months prior to enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) — http://www2.niddk.nih.gov/